CLINICAL TRIAL: NCT00736502
Title: Longterm Efficacy and Safety of NVP-based HAART in HIV-1 Positive Patients in the Daily Clinical Practice.
Brief Title: PMS Assessing the Long-term Efficacy and Safety of Nevirapine Therapy (Combined With Other ARV Drugs) in HIV-1 Positive Patients in Daily Clinical Practice.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1527
Record Dates: First submitted 2008-07-07; First posted 2008-08-18 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients HIV-1 positive

SUMMARY:
The aim of this trial is to evaluate the safety and virological and immunological efficacy of Viramune® on a background of different antiretroviral drug combinations.

ELIGIBILITY:
Inclusion criteria:

The inclusion criteria follow the same criteria which are describe in the newest SPC.

Exclusion criteria:

The exclusion criteria follow the same criteria which are describe in the newest SPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (17):
- Austria (7):
  - Boehringer Ingelheim Investigational Site 1, Graz
  - Boehringer Ingelheim Investigational Site 2, Linz
  - Boehringer Ingelheim Investigational Site 3, Salzburg
  - Boehringer Ingelheim Investigational Site 4, Vienna
  - Boehringer Ingelheim Investigational Site 5, Vienna
  - Boehringer Ingelheim Investigational Site 6, Vienna
  - Boehringer Ingelheim Investigational Site 7, Wels
- Poland (10):
  - Boehringer Ingelheim Investigational Site 8, Bialystok
  - Boehringer Ingelheim Investigational Site 9, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 10, Chorzów
  - Boehringer Ingelheim Investigational Site 11, Gdansk
  - Boehringer Ingelheim Investigational Site 12, Krakow
  - Boehringer Ingelheim Investigational Site 13, Lódz
  - Boehringer Ingelheim Investigational Site 14, Poznan
  - Boehringer Ingelheim Investigational Site 15, Szczecin
  - Boehringer Ingelheim Investigational Site 16, Warsaw
  - Boehringer Ingelheim Investigational Site 17, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 280 patients enrolled but two patients were lost to follow up before the second visit (2 weeks). For these two patients no information about Nevirapine intake could be assessed. So they were not included in the treated set which was used for most of the analyses.
Pre-assignment Details: This was an observational, non-interventional, uncontrolled, prospective post marketing study.
Groups:
- Nevirapine: Patients treated with 200 mg Nevirapine twice daily (administered orally).
Period: Overall Study
Arm/Group | Nevirapine
Started | 278 (Entered and treated.)
Completed | 213
Not Completed | 65
Not completed — Adverse Event | 22
Not completed — Lack of Efficacy | 16
Not completed — Lost to Follow-up | 27

BASELINE CHARACTERISTICS:
Population: Treated set
Arm/Group | Nevirapine
Number analyzed (Participants) | 278
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 219

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Reporting Adverse Events
Description: the incidence of non serious adverse events and serious adverse events according to body system (= System Organ Class) and preferred term.
Time Frame: 48 weeks
Population: The treated Set (TS), defined as all patients reported to have received at least one dose of Nevirapine.
Measure: Number; unit: Percentage of participants
Arm/Group | Nevirapine
Number analyzed (Participants) | 278
Percentage of participants
  any event | 25.5
  serious adverse events | 4.3
  adverse events leading to discontinuation | 9.7
  rash, any severity | 3.2
  hepatic events, any severity | 3.2
  Central Nervous system side effects, any severity | 3.6

2. Secondary Outcome: Virologic Response (VR)
Description: VR was defined as Human immunodeficiency virus (HIV) viral load of <50 copies/mL before week 48 and without any subsequent rebound or change of Antiretroviral (ARV) therapy. A rebound was defined by two consecutive measurements of Viral load (VL) >= 50 copies/mL, at least two weeks apart, after two consecutive measurements of VL < 50 copies/mL. A change of ARV therapy was defined as a permanent discontinuation of Nevirapine.
Time Frame: 48 weeks
Population: TS
Measure: Number; unit: Participants
Arm/Group | Nevirapine
Number analyzed (Participants) | 278
Participants
  with VR | 139
  without VR | 16
  missing | 123

3. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 48
Description: Calculated as CD4+ cell count at week 48 minus the baseline value
Time Frame: Baseline and week 48
Population: TS with non-missing data at baseline and week 48
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Nevirapine
Number analyzed (Participants) | 155
Cells/mm^3 | 148.5 (154.6)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Nevirapine
Serious Adverse Events (participants affected / at risk) | 12/278
Other Adverse Events (participants affected / at risk) | 0/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine (N=278)
Anemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy, generalised (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cholecystitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Malaise (General disorders) | 1
Pregnancy (General disorders) | 1
Clostridia enteritis (Infections and infestations) | 1
Helicobacter phylori infection (Infections and infestations) | 1
porta catheter infection (Infections and infestations) | 1
Staphylococcus sepsis (Infections and infestations) | 1
Fracture of foot (Injury, poisoning and procedural complications) | 1
Hyperkaliemia (Investigations) | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 1
Lymphoma of the brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes insipitus (Nervous system disorders) | 1
Pneumocystitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Enanthema (Skin and subcutaneous tissue disorders) | 1
Herpes eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Fever (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Pulmonary embolism (Vascular disorders) | 2
Shunt thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.